CLINICAL TRIAL: NCT04433273
Title: A Randomized, Double-blind, Sham-controlled Trial to Evaluate Changes in AMPK Following Daily Vestibular Nerve Stimulation (VeNS) in Adults Who Are Overweight or Obese.
Brief Title: Electrical Vestibular Stimulation (VeNS): Assessment of AMPK & SIRT1 Following Repeated Usage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: Compliance Solutions Ltd. (Industry); RD Gardi Medical College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVS002A
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Healthy control group (No Intervention): Neither placebo nor vestibular stimulation is administered
- Group B: Placebo control group (Placebo Comparator): Placebo stimulation along with regular treatment
  Interventions: Device: Electrical vestibular nerve stimulation
- Group C: Intervention group (Active Comparator): Electrical vestibular nerve stimulation along with regular treatment
  Interventions: Device: Electrical vestibular nerve stimulation

INTERVENTIONS:
Device: Electrical vestibular nerve stimulation — Electrical vestibular nerve stimulation using a headset device
  Arms: Group B: Placebo control group; Group C: Intervention group

SUMMARY:
The vestibular system which is responsible for balance and equilibrium constitutes our sixth sense. Metabolic Syndrome is a constellation of metabolic abnormalities characterized by obesity, insulin resistance (diabetes mellitus), hypertension, and dyslipidemia. It is generally agreed that a combination of three or more of the following components must be present: large waist circumference, elevated triglyceride, decreased high-density lipoprotein (HDL) cholesterol raised blood pressure, and elevated fasting blood sugar (FBS). Sirtuin 1 (SIRT1) is one of seven mammalian orthologs of the yeast protein silent information regulator. It is a conserved NAD-dependent protein deacetylase that decreases in cells that have high insulin resistance. In vivo, insulin resistance and metabolic syndrome were associated with low SIRT1 gene and protein expression. SIRT1 plays an important role to stimulate AMPK in improving mitochondrial function both in-vitro and in-vivo. Adenosine 5'-monophosphate (AMP)-activated protein kinase (AMPK) is a key factor in regulating energy metabolism, placing it at the center stage in studies of diabetes and related metabolic disorders like metabolic syndrome. It was reported that over a period of 6 weeks regular vestibular rehabilitation exercises caused an increase in the expression of SIRT1. The sleep inducing effects of vestibular stimulation is well known. Earlier studies reported improvement in the scores of Pittsburgh Sleep Quality Index (PSQI) and Epworth Sleepiness Scale (ESS) followed by the vestibular stimulation. Hence, we hypothesize that vestibular stimulation will lead to up-regulation of both SIRT1 and AMPK.

ELIGIBILITY:
Inclusion Criteria:

Male and female participants 35-60 years of age group Metabolic syndrome (BMI 25-35 kg/m2) Type 2 Diabetes Hyperlipidemia Willing participants

Exclusion Criteria:

Using Beta blockers Ear problems ( assessed during physical examination) Under any kind of therapy or treatment With severe complications Vestibular disorders

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of SIRT1 (Sirtuin 1) | 4 weeks
  SIRT1 (Sirtuin 1) levels will be assessed from the blood samples by ELISA method using respective kits.
AMPK | 4 weeks
  AMPK levels will be assessed from the blood samples by ELISA method using respective kits.

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 4 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a standard questionnaire used to assess sleep quality and quantity for the last month. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
  Minimum value = 0 Maximum value = 21
The Epworth Sleepiness Scale (ESS) | 4 weeks
  The Epworth Sleepiness Scale (ESS) is a standard questionnaire used as a subjective measure of a patient's sleepiness.
  Minimum value = 0 Maximum value = 24 A higher score indicates worse outcome (excessive sleepiness)

CONTACTS AND LOCATIONS:
Locations (1):
- RD Gardi Medical College, Ujjain, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: No
Data will be transferred in an encrypted PDF format. Trial staff will be given direction on how to share the trial data and given access to one specific section of a controlled cloud service which is controlled via role based access. Once they have authenticated with the service and the service verifies that they have the correct role to access the system they will be directed to a single webpage within the application where they will be able to upload the encrypted PDF. This PDF is generated on the fly and is therefore not stored in another location that could become compromised. Generating the PDF on the fly means that the source data is extracted from the database, processed and delivered in the context of a single request. These data will be transferred for each subject when they complete participation in the study.